CLINICAL TRIAL: NCT00088686
Title: Evaluation of Vanilloid Receptor Inactivation for Preemptive Analgesia
Brief Title: Capsaicin to Control Pain Following Third Molar Extraction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040248; 04-D-0248
Record Dates: First submitted 2004-07-30; First posted 2004-08-02 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-10

CONDITIONS: Healthy; Tooth Extraction
Keywords: Preemptive Analgesia; Vanilloid; Capsaicin; Acute Pain; Orofacial; Vanilloid Receptor (VR); Visual Analog Scale (VAS); Wisdom Teeth; Third Molar Extraction
MeSH Terms: conditions — Acute Pain | interventions — Capsaicin

INTERVENTIONS:
Drug: Capsaicin (Intramucosal Injection)

SUMMARY:
Capsaicin to Control Pain Following Third Molar Extraction

Summary: This study will test the effectiveness of the drug capsaicin in controlling pain after third molar (wisdom tooth) extraction. Capsaicin, the ingredient in chili peppers that makes them "hot," belongs to a class of drugs called vanilloids, which have been found to temporarily inactivate pain-sensing nerves. If capsaicin alleviates pain in dental surgery, it may have potential for use in many types of surgery and painful illnesses.

Healthy normal volunteers between 16 and 40 years of age who require third molar (wisdom tooth) extraction may be eligible for this study. Participants undergo the following procedures in three visits:

Visit 1

Patients have touch (sensory) testing inside the mouth using three methods: 1) applying a temperature probe onto the gums and having the patient rate how warm it is; 2) applying a gentle stroke across the gums with the bristles of a small paint brush and having the patient say whether or not it feels painful; and 3) applying a light touch to the gums with a small needle and having the patient rate the pain intensity following the touch. Following touch testing, the patient's mouth is numbed with an anesthetic and a small piece of gum tissue next to the lower wisdom tooth is removed (biopsied). Then, a small amount of either capsaicin or placebo (saline, or salt water) is injected next to the wisdom tooth.

Visit 2

Following repeat the touch testing, patients are sedated with an injection of midazolam. They then have another biopsy under local anesthesia on the same side of the mouth as the first biopsy. Their mouth is again numbed with an anesthetic, and they are given either a pain-relieving medicine called Toradol or a placebo injected into the arm. One lower wisdom tooth is then extracted. After the extraction, pain ratings are recorded every 20 minutes for up to 6 hours. During this time, patients are monitored for vital signs, numbness, pain, and side effects. Patients who request pain-relief medication are given acetaminophen and codeine. At the end of the study, they are discharged from the clinic and given acetaminophen and codeine to take at home, as instructed. They are provided a pain diary to record pain ratings and any adverse reactions that might occur until the last visit.

Visit 3

Patients return for a follow-up evaluation 48 hours after discharge from the clinic. At the end of the evaluation, they are discharged home with flurbiprofen for pain relief. Remaining wisdom teeth are removed "off-study" no sooner than 1 week following the first visit.

DETAILED DESCRIPTION:
Successful preemptive analgesic strategies are superior to traditional pain management schemes in the management of post-operative pain. The premise of this double-blind, placebo and positive-controlled clinical study is to evaluate the efficacy of vanilloid agonists as preemptive agents in an oral surgery tissue injury model. Vanilloids are a class of small organic compounds; the most familiar of which is capsaicin, the active ingredient in hot pepper. Binding of capsaicin to the vanilloid-1 receptor produces initial activation and then long-acting desensitization of pain specific neurons. We propose to produce a selective, long-term inactivation of peripheral pain transmission through the local application of capsaicin in the oral mucosa in an effort to prevent or reduce post-operative pain in the oral surgery model. Healthy subjects will be recruited, and following local anesthesia and conscious sedation, will be given an intramucosal injection of either capsaicin or placebo, or as a positive control, intravenous ketorolac. Subjects will rate pain and time of analgesic rescue medication request will be noted. Small biopsies will be removed from the extraction site prior to drug injection and at 48 hr post-operatively. Tissue levels of neurogenic inflammatory mediators and sensory neuron content will be compared pre- and post-operatively. A decrease in post-operative pain and decrease in analgesic use will be taken as a positive effect of the vanilloid for decreasing post-operative pain. We anticipate that through the long term blockade of pain specific fibers pre-operatively that there will be significant attenuation of post-operative pain development following surgery. This has significant implications for reducing pain and suffering, decreasing analgesic use, and reducing post-operative complications following surgery.

ELIGIBILITY:
INCLUSION CRITERIA:

Male or female volunteers referred for mandibular third molar extraction with a minimal difficulty rating score of 2 - 3 at the time of screening; rating will be verified by the oral surgeon at time of surgery. (Rating scale: 1 = erupted; 2 = soft tissue impaction; 3 = partial bony impaction; 4 = full bony impaction).

Age between 16-40.

ASA status 1 or 2, deemed in good general health (able to tolerate outpatient conscious sedation safely).

Willing to wait up to 4 hours for post-operative observation.

Willing to return at 48 hours for a second tissue biopsy.

EXCLUSION CRITERIA:

ASA status 3-5 and Emergency operation (E) that do not get a physician clearance; i.e. systemic disturbances that limits the patient's activity.

Pregnant or breast-feeding mothers.

Allergy to investigational drugs or to red chili peppers.

Chronic use of analgesics (not limited to, but including: non-steroidal anti-inflammatory medications, steroids, anti-depressants, anti-convulsants).

Presence of chronic disease (e.g. cardiovascular disease, liver disease, kidney disease, diabetes, etc.).

No exclusions will be made based on race, gender, or religion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75
Dates: Start 2004-07; Study Completion 2005-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Dental And Craniofacial Research (NIDCR), Bethesda, Maryland, United States

REFERENCES:
- [Background] Baranowski R, Lynn B, Pini A. The effects of locally applied capsaicin on conduction in cutaneous nerves in four mammalian species. Br J Pharmacol. 1986 Oct;89(2):267-76. doi: 10.1111/j.1476-5381.1986.tb10256.x. PMID 3779210
- [Background] Berger A, Henderson M, Nadoolman W, Duffy V, Cooper D, Saberski L, Bartoshuk L. Oral capsaicin provides temporary relief for oral mucositis pain secondary to chemotherapy/radiation therapy. J Pain Symptom Manage. 1995 Apr;10(3):243-8. doi: 10.1016/0885-3924(94)00130-D. PMID 7629418
- [Background] Bevan S, Szolcsanyi J. Sensory neuron-specific actions of capsaicin: mechanisms and applications. Trends Pharmacol Sci. 1990 Aug;11(8):330-3. doi: 10.1016/0165-6147(90)90237-3. PMID 2203194